CLINICAL TRIAL: NCT03190603
Title: Effects of Nonsteroidal Anti-inflammatory Drug (NSAID) on Inflammatory Lesion of Axial Spondyloarthritis Results From MRI Finding
Brief Title: Effects of Nonsteroidal Anti-inflammatory Drug (NSAID) on Inflammatory Lesion of Axial Spondyloarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Armed Forces Capital Hospital, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Hong Ki Min, M.D., Armed Forces Capital Hospital, Republic of Korea
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Hong Ki Min
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Spondylarthropathies; Magnetic Resonance Imaging
MeSH Terms: conditions — Spondylarthropathies | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Celecoxib arm (Experimental): Axial Spondyloarthritis patients who takes celecoxib 400mg for day
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — Continue celecoxib 400mg/day for 3months in axial spondyloarthritis patients.

SUMMARY:
Axial Spondyloarthritis (SpA) is a kind of inflammatory arthritis which includes ankylosing spondylitis. Common symptoms of axial SpA are inflammatory back pain, morning stiffness, peripheral arthritis, enthesitis. Controlling aforementioned symptoms are one of the goal in treatment, and another goal is preventing bony ankylosis of axial skeleton such as spine. Ankylosis can limit range of motion and lower the quality of life.

Non-steroidal antiinflammatory drug (NSAID) and Tumor necrosis factor (TNF)-a inhibitor are the current treatment options for axial SpA. These medications can improve pain and stiffness of axial SpA patients, however preventing bony ankylosis is not proven. Current study showed attenuating inflammation at early stage could prevent further bony destruction and ankylosis in axial SpA. Present study is designed to discover the therapeutic effect of NSAID whether NSAID could recover the early inflammatory bony change (bone marrow edema at MRI) and prevent further bony change.

ELIGIBILITY:
Inclusion Criteria:

1. 2009 Assessment of SpondyloArthritis international Society (ASAS) classification criteria for axial spondyloarthritis
2. Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) > 4
3. definite bone marrow edema on Sacroiliac joint MRI

Exclusion Criteria:

1. Patients who have underling cancer / infectious disease / kidney disease / liver disease / cardiovascular or cerebrovascular disease
2. Patients who is using TNF-a inhibitor
3. Patients with side effects of NSAID
4. Patients with history of peptic ulcer
5. Patients who can't keep NSAID treatment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Spondyloarthritis Research Consortium of Canada (SPARCC) MRI score of sacroiliac joint | Baseline, 6 weeks after, 12 weeks after
  Change from baseline SPARCC MRI score of sacroiliac joint at 6 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Capital Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No